CLINICAL TRIAL: NCT01801176
Title: Peripheral Primitive Fibromatosis. Study Evaluating a Simple Initial Monitoring With Search of Scalability Predictive Factors and Registration of Treatments in Case of Progression
Brief Title: Peripheral Primitive Fibromatosis
Acronym: WS-RT Fibro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2011-A01188-33; 2011/1774 (Other: CSET number)
Record Dates: First submitted 2013-02-25; First posted 2013-02-28 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Peripheral Primitive Fibromatosis
Keywords: proved by biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Initial monitoring group (Experimental)
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MRI every 3 months during the first year and then every 6 months during the second year and then one MRI up to 36 months

SUMMARY:
It's a monitoring study. The aim is to assess the progression free survival up to 3 years. Patients are not treated until progression. Search for scalability predictive factors and registration of treatments if progression.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral primitive fibromatosis
* Adults patients
* Peripheral primitive fibromatosis proved by biopsy
* Peripheral primitive fibromatosis R2 resected for which monitoring is decided
* MRI realized before inclusion
* Patient information and informed consent signed

Exclusion Criteria:

* Local recur
* Head and neck topography
* Primitive fibromatosis R0 or R1 resected
* Specific medical treatment of fibromatosis
* Patient already included in an other clinical trial with an experimental molecule
* Persons deprived of liberty
* Impossibility to submit to the trial's medical follow-up for psychological, geographical or socials reasons
* Previous history of cancer
* Counter indication to the realization of an MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | assessed up to 3 years

SECONDARY OUTCOMES:
Functional result | 1 year
  Assessed with criteria for Adverse Effects-V4 scale once per year during the consultation

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, Val de Marne, France